CLINICAL TRIAL: NCT07318311
Title: Comparative Evaluation of the Effect of pH Adjustment of the Solution of Articaine With Epinephrine on the Efficacy of Jet Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 0620152
Record Dates: First submitted 2025-12-23; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Comparative Evaluation of the Effect of pH Adjustment of the Solution of Articaine With Epinephrine on the Efficacy of Jet Anesthesia
Keywords: articaine, buffer, alkalization, needle-free local anesthesia, jet system
MeSH Terms: interventions — Anesthesia, Local; Carticaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control-Non buffered (Other): Local anesthesia administration articaine 4% with adrenaline 1/100000 via Comfort-in device
  Interventions: Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine by using Comfort-in device; Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine with the addition of sodium bicarbonate 8,4% by using Comfort-in device
- Experimental-buffered (Experimental): Local anesthesia administration articaine 4% with adrenaline 1/100000 with the addition of sodium bicarbonate 8,4% via Comfort-in device
  Interventions: Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine by using Comfort-in device; Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine with the addition of sodium bicarbonate 8,4% by using Comfort-in device

INTERVENTIONS:
Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine by using Comfort-in device — Implementation of local anesthesia with the usage of the jet device Comfort-In in the area of the upper central incisor of the right quadrant (#11). Specifically, the anesthetic solution infused was 0.3ml of articaine 4% with adrenaline 1/100000.
Other: Local anesthesia with articaine 4% with 1:100.000 epinephrine with the addition of sodium bicarbonate 8,4% by using Comfort-in device — Implementation of local anesthesia with the usage of the jet device Comfort-In in the area of the upper central incisor of the right quadrant (#11). Specifically, the anesthetic solution infused was 0.3ml of articaine 4% with adrenaline 1/100000 with the addition of the regulatory solution of sodium bicarbonate 8,4%.

SUMMARY:
The purpose of this study is to evaluate the effect of pH adjustment of the solution of articaine 4% with epinephrine 1:100.00, on the efficacy of anesthesia with the usage of a local anesthesia device that is needle-free (Comfort-In), and uses pressure implementation. An additional purpose of the study is to evaluate the efficacy of the device and its acceptance by the patients.

DETAILED DESCRIPTION:
In the present clinical research of the Dental School of the Aristotle University of Thessaloniki, there were forty-five healthy adult participants (ASA I) with no dental or other phobia, not being pregnant or going through breastfeeding process, with a record free of any allergies caused by local anaesthetics or the intake of suppressant substances of the central nervous system (CNS), and with an intact upper central incisor jaw #11 (viable, non-inflamed pulp tissue without rehabilitation). The participants took part in the study voluntarily, after being informed about the process through a special information sheet, and then signing a printed consent form. Medical and dental record was taken afterwards, which included questions about the volunteer's general experience concerning local anaesthesia, and also clinical examination was carried out to find out whether the volunteers qualify for research inclusion. The next step was the implementation of local anaesthesia with the usage of the jet device Comfort-In in the area of the upper central incisor of the right quadrant (#11), held in two separate sessions, the second one occurring at least one week after the first one. Specifically, the double blind method was used and the anaesthetic solutions infused randomly were 0.3ml of articaine 4% with adrenaline 1/100000 and 0.3ml of articaine 4% with adrenaline 1/100000 with the addition of the regulatory solution of sodium bicarbonate 8,4%. Right after the infusion of each anaesthetic solution and every 2 minutes, vitality tests of the pulp via an electric pulp-tester as well as tests of the sensitivity of the gums via the implication of cotton forceps were held and recorded, until anaesthesia had gone away completely. During the session, while infusing the anaesthetic, an evaluation of the pain was held (visual, numerical and operational proportional scale of pain - VAS), and also, the participant replied to 6 questions by completing a corresponding questionnaire relevant to the acceptance of the technique. After 48 hours, the main researcher contacted every volunteer to record any post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy adults (ASA I) whose medical history allows the administration of local anesthesia with vasoconstrictor, 2) Volunteers without dental fear or any other phobia, 3) Volunteers males/females aged 18-35, 4) Volunteers with intact upper central incisor (#11) with viable, non-inflamed pulp tissue, without trauma history, periodontal disease, or decay, without rehabilitation.

Exclusion Criteria:

1) Allergy history in local anesthetic solutions, 2) Pregnancy or breastfeeding, 3) Pathological lesions or active inflammation spots in the area of infusion, 4) Volunteers that receive chronic medication that presents interactions with local anesthesia solutions and mainly with vasoconstrictors (e.g. TCA or b-blockers), and volunteers that have received suppressants of CNS up to 48 hours before the administration (e.g. alcohol or NSAIDs) as they cause disorder of sensibility.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-07 (Actual)

PRIMARY OUTCOMES:
Success rate of pulpal anesthesia | 2 minutes after the infusion of the anesthetic via Comfort-in
  Calculation of the percentage of participants with successful anesthesia via pulp-tester

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Dabarakis, Associate Professor, Study Chair — Aristotle University Of Thessaloniki; Theodoros Lilis, Assistant Professor, Study Director — Aristotle University Of Thessaloniki; Vasileios Kyros, Postgraduate Student, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Dental School Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manta K, Dabarakis N, Lillis T, Fotopoulos I. Anesthetic efficacy of buffered 4% articaine for mandibular first molar infiltration: a crossover clinical trial. J Dent Anesth Pain Med. 2023 Jun;23(3):135-141. doi: 10.17245/jdapm.2023.23.3.135. Epub 2023 May 26. PMID 37313270